CLINICAL TRIAL: NCT05212311
Title: Effect of Chitosan Phonophoresis On Cubital Tunnel Syndrome: A Randomized Controlled Trial
Brief Title: Effect of Chitosan Phonophoresis On Cubital Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy Ali Hassan ElMeligie, Principal investigator, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CUTS001
Record Dates: First submitted 2022-01-15; First posted 2022-01-28 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Cubital Tunnel Syndrome; Ulnar Nerve Entrapment at Elbow; Ulnar Nerve Compression; Ulnar Nerve Entrapment Syndrome
MeSH Terms: conditions — Cubital Tunnel Syndrome; Ulnar Nerve Compression Syndromes | interventions — Ultrasonic Therapy; Splints

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Control group) (Active Comparator): Group A (n=27) will receive a conventional physical therapy program only for 5 weeks in the form of Splinting, Ultrasound and Exercises.
  Interventions: Device: Chitosan Phonophoresis; Device: Splinting; Other: Neural mobilization exercises of the ulnar nerve
- Group B (Chitosan phonophoresis group) (Experimental): Patients in group B (n=27) will receive phonophoresis with chitosan nanoparticles. Patients will also receive the conventional physical therapy program: in the form of Splinting, Ultrasound and Exercises. Session will be applied 3 times per week for a total of 5 weeks.
  Interventions: Device: Therapeutic Ultrasound; Device: Splinting; Other: Neural mobilization exercises of the ulnar nerve

INTERVENTIONS:
Device: Chitosan Phonophoresis — Therapeutic pulsed ultrasound using EMS physio Ltd ultrasound device in presence of chitosan gel will be applied over the elbow. The following parameters will be used: US treatment was applied for 5 min per session at a frequency of 3 MHz and an intensity of 0.5 W/cm2 in pulsed mode with a transducer area of 5 cm2.
  Arms: Group A (Control group)
Device: Therapeutic Ultrasound — US treatment will be applied for 5 min per session at a frequency of 3 MHz and an intensity of 0.5 W/cm2 in pulsed mode with a transducer area of 5 cm2 using aquasonic gel.
  Arms: Group B (Chitosan phonophoresis group)
Device: Splinting — Splinting the elbow in comfortable flexion (40-70), forearm and wrist in neutral (slight forearm pronation and wrist flexion if symptoms are severe), can allow the nerve and surrounding supporting structures the rest and relief from compression and traction.
  The elbow portion of the splint should be well padded or ''bubbled out'' to provide pressure relief for the area of the cubital tunnel. It may be necessary to splint the ulnar digits of the hand to prevent contracture, maintain passive and active range of motion, and improve hand function. If the motor branch of the nerve is sufficiently involved to cause muscle denervation, a hand-based intrinsic plus splint or the use of finger-based splints to prevent clawing of the ring and small fingers will provide balanced positioning of the affected structures.
Other: Neural mobilization exercises of the ulnar nerve — Nerve mobilization exercises Inflammation or adhesions anywhere along the ulnar nerve path can cause the nerve to have limited mobility and essentially get stuck in one place. These exercises help stretch the ulnar nerve and encourage movement through the cubital tunnel

SUMMARY:
- This study will be conducted to answer the following question: Is there a statistically significant effect of chitosan phonophoresis on ulnar nerve conduction velocity, pain level & function in patients with mild to moderate cubital tunnel syndrome?

- Fifty-four subjects suffering from mild to moderate cubital tunnel syndrome according to modified McGowan grading system (Palmer & Hughes, 2010) from both sexes diagnosed clinically by electromyography will be recruited for this study. The Age of the participants will range from 20 - 40 years old. Participants with Body mass index between 18.5 and 24.9kg/m2.

EMS physio Ltd ultrasound device will be used in combination with chitosan nanoparticles gel.

Electrodiagnostic test will be performed for ulnar nerve conduction velocity using Neuropack S1 MEB-9004 NIHON KODEN, JAPAN. Visual analogue scale (VAS) will be used to determine pain level. Quick DASH will be used to determine hand function.Patients will have 3 sessions per week for 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Fifty-four patients suffering from mild to moderate Cubital tunnel syndrome from both sexes according to modified McGowan grading system (Palmer & Hughes, 2010) & have motor conduction velocity across the elbow less than 50 m/s or the difference between the motor conduction velocity across the elbow and that below the elbow exceeds 10 m/s (Padua et al., 2001).
2. Age ranging from 20-35.
3. All participants will have Body mass index between 18.5 and 24.9 kg/m2.

Exclusion Criteria:

* 1- Diabetic patients. 2- Cardiovascular patients 3- Patients with cervical spondylosis 4- Patients with cervical disc prolapsed 5- Patients with Thoracic outlet syndrome 6- Patients with carpal tunnel syndrome. 7- Pregnant women 8- Patients with fibromyalgia 9- Patients with epicondylitis 10- Patient with previous elbow injuries 11- Patient with Breast Cancer. 12- Patient with Guyon Canal syndrome 13- Smokers

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Changes in ulnar nerve conduction velocity from baseline and 5 weeks posttreatment | Changes in ulnar nerve conduction velocity from baseline and 5 weeks posttreatment
  Measurement of how quickly an electrical impulse moves along the nerve.

SECONDARY OUTCOMES:
Changes in pain intensity at 5 weeks posttreatment | Changes in pain intensity from baseline and 5 weeks posttreatment
  pain (min-max:0-10) Higher scores correlate to higher intensity of pain
Changes in function using QUICK DASH scale at 5 weeks posttreatment | Changes in function using QUICK DASH scale from baseline and 5 weeks posttreatment
  the quickdash is a validated outcome measure for hand function, scored 0-100 with higher scores indicating worse disability which is bad.

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 University Hospital, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all of the individual participant data collected during the trial and after deidentification
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 Months after study publication
Access Criteria: Email: mohamed.magdy.pt@o6u.edu.eg